CLINICAL TRIAL: NCT02352753
Title: To Evaluate the Effect of Denosumab in Lumbar Spine Bone Mineral Density (BMD) Z-score at 12 Months, as Assessed by Dual-energy X-ray Absorptiometry (DXA), in Children 2 to 17 Years of Age (at the Time of Screening) on a 3-Month Dosing Regimen With OI
Brief Title: Multicenter,Single-arm Study to Evaluate Efficacy, Safety, & Pharmacokinetics of Denosumab in Children w/ OI
Acronym: OI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped earlier than planned due to safety concerns about high levels of calcium in the blood of the participants
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20130173; 2014-000184-40 (EudraCT Number)
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Osteogenesis Imperfecta
Keywords: Amgen, OI, Bone
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Denosumab (Experimental): Participants received denosumab 1 mg/kg (up to a maximum of 60 mg) subcutaneously every 6 months (Q6M) for up to 36 months.
  Early efficacy and PK data from Q6M dosing supported adjustment of the dosing regimen from Q6M to every 3 months (Q3M). Participants enrolled and still receiving denosumab were transitioned from Q6M to Q3M dosing schedule. Participants could transition to Q3M dosing schedule up to and including the date they attended for their month 36 visit under the Q6M dosing regimen. Those participants received denosumab during the Q3M dosing regimen for 12 months. Participants who transition to Q3M at month 18 of the Q6M dosing regimen received denosumab Q3M for up to 18 months.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Subcutaneous (SC) injection.

SUMMARY:
This is a prospective, multicenter, single-arm study in children 2 to 17 years of age with OI to evaluate efficacy and safety of denosumab.

DETAILED DESCRIPTION:
To evaluate the effect of denosumab in lumbar spine bone mineral density (BMD) Z-score at 12 months, as assessed by dual-energy X-ray absorptiometry (DXA), in children 2 to 17 years of age (at the time of screening) on a 3-Month Dosing Regimen with osteogenesis imperfecta (OI)

ELIGIBILITY:
• Eligibility criteria relates to initial enrollment into this study (6-Month Dosing Regimen). Subjects reconsenting to a 3-Month Dosing Regimen will not repeat eligibility assessments

Inclusion Criteria:

• Clinical diagnosis of OI defined as a clinical history consistent with type I-IV OI Clinical severity of OI as defined by 2 or more prevalent vertebral compression fractures; OR1 prevalent vertebral compression fracture and 1 or more nonvertebral fractures within the previous 2 years; OR 3 or more fractures within the previous 2 years.

Exclusion Criteria:

* Inability or unwillingness to comply with the requirements for frequent calcium and phosphorus monitoring for 14 days after the first dose of denosumab (only applies to the first 5 subjects age 11 to17 enrolled in the study and the first 5 subjects of any age meeting the criteria for increased bone turnover
* Currently unhealed fracture or osteotomy as defined by orthopedic opinion
* Osteotomy within 5 months of screening
* Evidence of untreated oral cavities or oral infections
* Recent or planned invasive dental procedure
* Surgical tooth extraction which has not healed by screening
* History of an electrophoresis pattern inconsistent with type I to IV OI
* History of genetic testing results inconsistent with type I to IV OI
* Abnormalities of the following per central laboratory reference ranges at screening: Serum albumin corrected calcium < lower limit of normal (LLN) Serum vitamin D < 20 ng/mL; re-screening for Vitamin D level < 20 ng/mL will be allowed, after adequate supplementation
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 1.5 x upper limit of normal (ULN)
* Total bilirubin (TBL) > 1.5 x ULN (subjects with Gilbert syndrome are eligible)
* Serum phosphorus < LLN
* Serum alkaline phosphatase > 20% above the ULN or > 20% below the LLN
* Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 (calculated bythe Schwartz equation at screening) Evidence of any of the following: Current hyperthyroidism (unless well-controlled on stable antithyroid therapy)
* Current clinical hypothyroidism (unless well-controlled on stable thyroid replacement therapy)
* History of hyperparathyroidism
* Current hypoparathyroidism
* Current, uncontrolled hypercalcemia (albumin-corrected serum Ca >10% ULN)
* History of osteomalacia or rickets (chart review)
* Other bone diseases that affect bone metabolism (eg, osteoporosis pseudoglioma syndrome, idiopathic juvenile osteoporosis, osteopetrosis, hypophosphatasia)
* History of autoimmune disease
* History of rare hereditary problems of fructose intolerance
* Positive blood screen for human immunodeficiency virus -1 or -2 antibody
* Positive blood screen for hepatitis B surface antigen or hepatitis C antibody
* Received other osteoporosis treatment or bone active treatment with the following guidelines:
* Prior treatment with

  * denosumab
  * fluoride or strontium for bone disease (fluoride taken for routine dental care is permitted)
  * parathyroid hormone (PTH) or PTH derivatives within 12 months prior to screening
  * zoledronic acid within 6 months prior to screening
  * oral bisphosphonates or intravenous bisphosphonates other than zoledronic acid if the first dose of denosumab would be before their next scheduled bisphosphonate dose would have been given
* Administration of systemic glucocorticoids (≥ 5.0 mg prednisone equivalents/day for more than 10 days) within 3 months of screening.
* Topical and inhaled glucocorticoids will be allowed
* Administration of any of the following treatment within 3 months of screening:

  * Growth hormone (subjects on stable dose of growth hormone for at least 3 months prior to screening will be allowed)
* Currently receiving treatment in another investigational drug study, or less than 30 days since ending treatment on another investigational drugstudy(s), or current or planned participation in a clinical trial that would preclude compliance with study requirements Other inclusion/exclusion criteria may apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (47):
- United States (13):
  - Research Site, Los Angeles, California
  - Research Site, Torrance, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Decatur, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Omaha, Nebraska
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Australia (2):
  - Research Site, Westmead, New South Wales
  - Research Site, Subiaco, Western Australia
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Bulgaria (2):
  - Research Site, Sofia
  - Research Site, Varna
- Canada (3):
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (5):
  - Research Site, Hradec Králové
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Zlín
- France (4):
  - Research Site, Bordeaux
  - Research Site, Paris
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Toulouse
- Research Site, Cologne, Germany
- Research Site, Budapest, Hungary
- Italy (2):
  - Research Site, Roma
  - Research Site, Verona
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Lodz
  - Research Site, Rzeszów
  - Research Site, Warsaw
- Spain (3):
  - Research Site, Esplugues de Llobregat, Catalonia
  - Research Site, Getafe, Madrid
  - Research Site, Valencia, Valencia
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Bristol
  - Research Site, Glasgow
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 32 centers in North America, Europe, and Australia from June 2015 to March 2022.
Groups:
- Denosumab: Participants received denosumab 1 mg/kg (up to a maximum of 60 mg) subcutaneously every 6 months (Q6M) for up to 36 months.
  Participants were dose adjusted from Q6M to every 3 months (Q3M) after early efficacy and pharmacokinetic (PK) data were analyzed. Participants enrolled and still receiving denosumab were transitioned from Q6M to Q3M dosing schedule. Participants could transition to Q3M dosing schedule up to and including the date they attended for their Month 36 visit under the Q6M dosing regimen. Those participants received denosumab during the Q3M dosing regimen for 12 months. Participants who transitioned to Q3M at month 18 of the Q6M dosing regimen received denosumab Q3M for up to 18 months.
Period: 6-Month Dosing Period
Arm/Group | Denosumab
Started | 153
Received Investigational Product | 153
Completed | 55
Not Completed | 98
Not completed — Decision by sponsor | 2
Not completed — Withdrawal by Subject | 34
Not completed — Lost to Follow-up | 2
Not completed — Transitioning to Q3M | 60
Period: 3-Month Dosing Period
Arm/Group | Denosumab
Started | 60
Received Investigational Product | 60
Completed | 40
Not Completed | 20
Not completed — Decision by sponsor | 14
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who enrolled into the study.
Groups:
- Denosumab: Participants received denosumab 1 mg/kg (up to a maximum of 60 mg) subcutaneously every 6 months (Q6M) for up to 36 months.
  Participants were dose adjusted from Q6M to every 3 months (Q3M) after early efficacy and PK data were analyzed. Participants enrolled and still receiving denosumab were transitioned from Q6M to Q3M dosing schedule. Participants could transition to Q3M dosing schedule up to and including the date they attended for their Month 36 visit under the Q6M dosing regimen. Those participants received denosumab during the Q3M dosing regimen for 12 months. Participants who transitioned to Q3M at month 18 of the Q6M dosing regimen received denosumab Q3M for up to 18 months.
Arm/Group | Denosumab
Number analyzed (Participants) | 153
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data presented is the age at Q6M dosing regimen enrolment.
  Years | 9.3 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 138
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Black or African American | 2
  White | 135
  Other | 8
  Multiple | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) Z-Score at 12 Months
Description: Lumbar spine BMD was measured by dual-energy X-ray absorptiometry (DXA) adjusted for age, sex, and race/ethnicity. The results were then converted to Z-scores. The Z-score indicated the number of standard deviations away from the reference population and a score of 0 is equal to the mean. Positive changes from Baseline indicated an improvement in lumbar spine BMD.
Time Frame: Baseline and 12 months
Population: DXA Analysis Set included all participants in the FAS with Baseline and Month 12 DXA assessment on the Q3M dosing regimen for lumbar spine as provided by the central imaging vendor.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Groups:
- Denosumab 3-Month Dosing Regimen: Participants were dose adjusted from Q6M to every 3 months (Q3M) after early efficacy and PK data were analyzed. Participants enrolled and still receiving denosumab were transitioned from Q6M to Q3M dosing schedule. Participants could transition to Q3M dosing schedule up to and including the date they attended for their Month 36 visit under the Q6M dosing regimen. Those participants received denosumab during the Q3M dosing regimen for 12 months. Participants who transitioned to Q3M at month 18 of the Q6M dosing regimen received denosumab Q3M for up to 18 months.
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 45
Z-score | 1.009 (0.119)

2. Secondary Outcome: Change From Baseline in Lumbar Spine BMD Z-score at 6 Months
Description: Lumbar spine BMD was measured by DXA adjusted for age, sex, and race/ethnicity. The results were then converted to Z-scores. The Z-score indicated the number of standard deviations away from the reference population and a score of 0 is equal to the mean. Positive changes from Baseline indicated an improvement in lumbar spine BMD.
Time Frame: Baseline and 6 months
Population: DXA Analysis Set included all participants in the FAS with Baseline and Month 6 DXA assessment on the Q3M dosing regimen for lumbar spine as provided by the central imaging vendor.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Groups:
- Denosumab 3-Month Dosing Regimen: Participants were dose adjusted from Q6M to every 3 months (Q3M) after early efficacy and PK data were analyzed. Participants enrolled and still receiving denosumab were transitioned from Q6M to Q3M dosing schedule. Participants could transition to Q3M dosing schedule up to and including the date they attended for their month 36 visit under the Q6M dosing regimen. Those participants received denosumab during the Q3M dosing regimen for 12 months. Participants who transition to Q3M at month 18 of the Q6M dosing regimen received denosumab Q3M for up to 18 months.
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 54
Z-score | 0.925 (0.078)

3. Secondary Outcome: Change From Baseline in Proximal Femur BMD Z-score at 6 and 12 Months
Description: Proximal femur (total hip and femoral neck) BMD Z-score was measured by DXA adjusted for age, sex, and race/ethnicity. The results were then converted to Z-scores. The Z-score indicated the number of standard deviations away from the reference population and a score of 0 is equal to the mean. Positive changes from Baseline indicated an improvement in lumbar spine BMD.
Time Frame: Baseline, 6 and 12 months
Population: DXA Analysis Set included all participants in the FAS with Baseline, Month 6 and Month 12 DXA assessment on the Q3M dosing regimen for lumbar spine as provided by the central imaging vendor. Only participants 5 years of age or older are included.
Measure: Least Squares Mean (Standard Error); unit: Z score
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 32
Z score
  Total hip BMD Z-score - 6 Months | 0.799 (0.082)
  Total hip BMD Z-score - 12 Months | 0.793 (0.154)
  Femoral neck BMD Z-score - 6 Months | 0.769 (0.067)
  Femoral neck BMD Z-score - 12 Months | 0.689 (0.131)

4. Secondary Outcome: Percentage of Participants With at Least 1 X-ray Confirmed Long Bone or New and Worsening Vertebral Fracture
Time Frame: Q6M Dosing Regimen: Last 12 months of treatment (median treatment duration was 730.0 days); Q3M Dosing Regimen: Day 1 up to 12 months
Population: Q3M Dosing Regimen Safety Analysis Set: includes all participants in the FAS who received ≥ 1 dose of Q3M dosing regimen.
Measure: Number; unit: Percentage of participants
Groups:
- Denosumab 6-Month Dosing Regimen: Participants received denosumab 1 mg/kg (up to a maximum of 60 mg) subcutaneously every 6 months (Q6M) for up to 36 months.
Arm/Group | Denosumab 6-Month Dosing Regimen | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 60 | 60
Percentage of participants | 28.3 | 26.7

5. Secondary Outcome: Percentage of Participants With at Least 1 X-ray Confirmed New and Worsening Vertebral Fracture
Time Frame: as for outcome 4
Population: The Vertebral Fracture Analysis Set: includes all participants in the FAS who had a readable non-missing baseline and ≥1 non-missing postbaseline X-ray vertebral evaluation on the Q3M dosing regimen as provided by the central imaging vendor.
Measure: Number; unit: Percentage of participants
Arm/Group | Denosumab 6-Month Dosing Regimen | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 47 | 47
Percentage of participants | 12.8 | 8.5

6. Secondary Outcome: Percentage of Participants With at Least 1 X-ray Confirmed New Vertebral Fracture
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Denosumab 6-Month Dosing Regimen | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 47 | 47
Percentage of participants | 10.6 | 6.4

7. Secondary Outcome: Percentage of Participants Wth at Least 1 X-ray Confirmed Improving Vertebral Fracture
Time Frame: Q3M Dosing Regimen: Baseline up to 12 months
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 47
Percentage of participants | 27.7

8. Secondary Outcome: Percentage of Participants With at Least 1 Vertebral and Nonvertebral Fracture
Time Frame: as for outcome 4
Population: Q3M Dosing Regimen Safety Analysis Set: includes all participants in the FAS who received ≥ 1 dose of Q3M dosing regimen. Only participants 5 years of age or older are included.
Measure: Number; unit: Percentage of participants
Arm/Group | Denosumab 6-Month Dosing Regimen | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 56 | 56
Percentage of participants | 28.6 | 30.4

9. Secondary Outcome: Change From Baseline in Child Health Questionnaire-Parent Form Physical Summary Score (CHQ-PF-50) at 12 Months
Description: The CHQ-PF-50 was a 50-item questionnaire completed by the parents or guardians of children between 5 and 18 years of age. The 50 questions measure 14 domains which were summarized as the physical and psychological summary scores. Each summary score was transformed and could range from 0 to 100, with higher score indicating better physical and psychosocial health. A negative change from Baseline indicates decreased well-being.
Time Frame: Baseline and 12 months
Population: Patient Reported Outcomes (PRO) Analysis Set: includes all participants in the FAS who had a baseline and ≥ 1 postbaseline valid PRO response on Q3M dosing regimen for the CHQ-PF-50. The CHQ-PF-50 analysis set only includes participants 5 years of age and older at screening.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 45
Score on a scale | -0.98 (15.41)

10. Secondary Outcome: Change From Baseline in CHQ-PF-50 Psychological Summary Score at 12 Months
Description: The CHQ-PF-50 was a 50-item questionnaire completed by the parents or guardians of children between 5 and 18 years of age. The 50 questions measure 14 domains which were summarized as the physical and psychological summary scores. Each summary score was transformed and could range from 0 to 100, with higher score indicating better physical and psychosocial health. A positive change from Baseline indicates improved well-being.
Time Frame: Baseline and 12 months
Population: PRO Analysis Set includes all participants in the FAS who had a baseline and ≥ 1 postbaseline valid PRO response on Q3M dosing regimen for the CHQ-PF-50. The CHQ-PF-50 analysis set only includes participants 5 years of age and older at screening
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 45
Score on a scale | 0.85 (8.57)

11. Secondary Outcome: Change From Baseline in Childhood Health Assessment Questionnaire (CHAQ) Disability Index Score at 12 Months
Description: The disability domain (questions 1-54) of the CHAQ was used to measure the participant's assessment of physical functioning or the parent's assessment of the child's physical functioning. The disability index comprised of 8 categories (dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and activities). Scoring ranged from 1 to 5; 1 was "without any difficulty," 2 was "with some difficulty," 3 was "with much difficulty," and 4 was "unable to do." An answer of "not applicable" was scored as a 5, but was not counted. If a child required assistance from another person or used an aid or other device for any of the 8 categories, the minimum score for that category was recorded as a 3. The CHAQ questions were scored and converted to a total index score ranging from 0 to 3. Negative change from Baseline indicates an improvement.
Time Frame: Baseline and 12 months
Population: PRO Analysis Set includes all participants in the FAS who had a baseline and ≥ 1 postbaseline valid PRO response on Q3M dosing regimen for the CHAQ disability index score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 51
Score on a scale | -0.06 (0.46)

12. Secondary Outcome: Change From Baseline in Wong-Baker Faces Pain Rating Scale (WBFPRS) at 12 Months
Description: Participants were asked to report their level of pain by choosing a face that best described their own pain (the corresponding number: 0, 2, 4, 6, 8, 10) were then recorded. The WBFPRS ranged from 0, "no hurt," to 10, "hurts worst". A negative change from baseline indicates an improvement.
Time Frame: Baseline and 12 months
Population: Patient Reported Outcomes (PRO) Analysis Set: includes all participants in the FAS who had a baseline and ≥ 1 postbaseline valid PRO response on Q3M dosing regimen for the WBFPRS.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 49
Score on a scale | 0.0 (1.7)

13. Secondary Outcome: Serum Concentration of Denosumab
Time Frame: Days 1 (predose), 10, 30, and 60, & weeks 12, 24, 36, 48, 60, 72 (end of study visit), early termination visit, & follow-up visit 12 weeks after last dose (average duration of treatment: 231 days)
Population: PK Analysis Set includes all participants in the 3QM dosing regimen safety analysis set who had ≥ 1 serum denosumab reported result on 3QM dosing regimen at any 1 time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 60
ng/mL
  Day 1: number analyzed (Participants) | 59
  Day 1 | 8.1 (62.0)
  Day 10: number analyzed (Participants) | 52
  Day 10 | 6685.4 (1761.8)
  Day 30: number analyzed (Participants) | 52
  Day 30 | 3840.5 (1329.9)
  Day 60: number analyzed (Participants) | 51
  Day 60 | 1291.4 (971.2)
  Week 12 Day 1: number analyzed (Participants) | 55
  Week 12 Day 1 | 406.2 (627.0)
  Week 24 Day 1: number analyzed (Participants) | 56
  Week 24 Day 1 | 589.8 (804.3)
  Week 36: number analyzed (Participants) | 52
  Week 36 | 835.1 (983.5)
  Week 48: number analyzed (Participants) | 49
  Week 48 | 647.3 (875.1)
  Week 60: number analyzed (Participants) | 3
  Week 60 | 1266.7 (861.1)
  Week 72: number analyzed (Participants) | 2
  Week 72 | 970.0 (1371.8)
  Early Termination Visit: number analyzed (Participants) | 8
  Early Termination Visit | 4.2 (11.8)
  Week 12 Follow-up Visit: number analyzed (Participants) | 5
  Week 12 Follow-up Visit | 72.6 (103.9)

14. Secondary Outcome: Serum Bone Turnover Marker (BTM) - Serum Type I Collagen C Telopeptide
Time Frame: Baseline and Days 10 and 30, and Months 3, 6, 9, 12, 15 and 18
Population: BTM Analysis Set: includes all participants in the 3QM dosing regimen safety analysis set who had baseline and ≥ 1 postbaseline assessment for the BTM endpoint of interest on Q3M dosing regimen.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 54
ng/L
  Baseline | 1136.5 (569.7)
  Day 10: number analyzed (Participants) | 50
  Day 10 | 174.4 (64.7)
  Day 30: number analyzed (Participants) | 48
  Day 30 | 176.5 (87.9)
  Month 3: number analyzed (Participants) | 50
  Month 3 | 498.4 (332.0)
  Month 6: number analyzed (Participants) | 49
  Month 6 | 537.1 (427.1)
  Month 9: number analyzed (Participants) | 48
  Month 9 | 539.0 (425.0)
  Month 12: number analyzed (Participants) | 42
  Month 12 | 681.2 (563.1)
  Month 15: number analyzed (Participants) | 13
  Month 15 | 1050.8 (758.8)
  Month 18: number analyzed (Participants) | 1
  Month 18 | 1290.0 (NA) — Evaluable samples were too low to calculated standard deviation.

15. Secondary Outcome: BTM - Bone-specific Alkaline Phosphatase (BSAP)
Time Frame: Baseline and Days 10 and 30, and Months 3, 6, 9, 12, and 15
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 59
μg/L
  Baseline | 69.22 (34.26)
  Day 10: number analyzed (Participants) | 56
  Day 10 | 70.88 (32.77)
  Day 30: number analyzed (Participants) | 53
  Day 30 | 56.28 (28.32)
  Month 3: number analyzed (Participants) | 57
  Month 3 | 498.4 (332.0)
  Month 6: number analyzed (Participants) | 54
  Month 6 | 40.30 (22.58)
  Month 9: number analyzed (Participants) | 55
  Month 9 | 51.17 (106.27)
  Month 12: number analyzed (Participants) | 47
  Month 12 | 40.02 (27.64)
  Month 15: number analyzed (Participants) | 14
  Month 15 | 49.49 (31.20)

16. Secondary Outcome: Change From Baseline in Growth Velocity at 12 Months
Description: Change from baseline in growth velocity was determined by calculating age-adjusted Z-scores for height, weight and body mass index (BMI).
  Height-for-age Z-score was defined as the difference between the participant's height and the median height for the population with the same age and gender, divided by the population standard deviation.
  The definitions of growth velocity based on weight and BMI were analogously calculated. To programmatically calculate the Z-scores, the National Center for Health Statistics percentiles growth charts, based on the 2000 Center for Disease Control and Prevention (CDC) (http://www.cdc.gov/growthcharts/c c_charts.htm), and the CDC Anthropometric Software Package 3.0 Z-scores were used.
  During normal growth, the change in z-score for each of the three should equal 0. A positive change in any of the three indicates growth acceleration, whereas a negative change indicates deceleration.
Time Frame: Baseline and 12 months
Population: Growth Velocity Analysis Set includes all participants in the FAS with non-missing height, weight, or BMI, as applicable, at Baseline and postbaseline on the Q3M dosing regimen. Only participants with observed data at Baseline and Month 12 are included.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Denosumab 3-Month Dosing Regimen
Number analyzed (Participants) | 48
Z-score
  Height -for-age Z-score | -0.01 (0.43)
  Weight-for-age Z-score | 0.01 (0.53)
  BMI-for-age Z-score | -0.07 (0.52)

ADVERSE EVENTS:
Time Frame: 6QM dosing regimen: Day 1 up to 36 months 3QM dosing regimen: Day 1 up to 24 weeks after last dose (median duration of treatment was 253 days)
Description: Q6M: The Q6M regimen safety analysis set included all participants in the FAS who received ≥ 1 dose of investigational product.
  Q3M: The Q3M regimen safety analysis set included all participants in the FAS who received ≥ 1 dose of investigational product.
Arm/Group | Denosumab 6-Month Dosing Regimen | Denosumab 3-Month Dosing Regimen
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/60
Serious Adverse Events (participants affected / at risk) | 52/153 | 12/60
Other Adverse Events (participants affected / at risk) | 141/153 | 38/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 6-Month Dosing Regimen (N=153) | Denosumab 3-Month Dosing Regimen (N=60)
Right ventricular dilatation (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Procedural failure (General disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 15 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 7 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 8 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 5 | 0
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 5 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 10 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 4 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device dislocation (Product Issues) | 4 | 0
Device failure (Product Issues) | 1 | 0
Device loosening (Product Issues) | 1 | 0
Adnexal torsion (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 6-Month Dosing Regimen (N=153) | Denosumab 3-Month Dosing Regimen (N=60)
Abdominal pain (Gastrointestinal disorders) | 13 | 0
Abdominal pain upper (Gastrointestinal disorders) | 9 | 2
Dental caries (Gastrointestinal disorders) | 9 | 1
Vomiting (Gastrointestinal disorders) | 13 | 2
Pain (General disorders) | 12 | 2
Pyrexia (General disorders) | 18 | 1
Gastroenteritis (Infections and infestations) | 8 | 0
Influenza (Infections and infestations) | 13 | 0
Nasopharyngitis (Infections and infestations) | 23 | 7
Upper respiratory tract infection (Infections and infestations) | 9 | 1
Contusion (Injury, poisoning and procedural complications) | 16 | 0
Fall (Injury, poisoning and procedural complications) | 25 | 6
Femur fracture (Injury, poisoning and procedural complications) | 16 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 8 | 3
Foot fracture (Injury, poisoning and procedural complications) | 16 | 2
Hand fracture (Injury, poisoning and procedural complications) | 15 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 12 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 12 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 11 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 6 | 3
Radius fracture (Injury, poisoning and procedural complications) | 14 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 10 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 17 | 3
Ulna fracture (Injury, poisoning and procedural complications) | 16 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 28 | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 50 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 57 | 11
Headache (Nervous system disorders) | 21 | 4
Hypercalciuria (Renal and urinary disorders) | 49 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02352753/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT02352753/SAP_001.pdf